CLINICAL TRIAL: NCT04190433
Title: AuTophagy Activation for Cardiomyopathy Due to Anthracycline tReatment (ATACAR) Trial
Brief Title: Autophagy Activation for the Alleviation of Cardiomyopathy Symptoms After Anthracycline Treatment, ATACAR Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively closed due to low/no accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-007547; NCI-2021-13928 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Breast Carcinoma; Hematopoietic and Lymphoid Cell Neoplasm; Lymphoma; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Hematologic Neoplasms; Lymphoma; Sarcoma | interventions — Carvedilol; Lisinopril; Pravastatin; Spironolactone; Acetates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (carvedilol, lisinopril) (Active Comparator): Patients receive carvedilol orally (PO) and lisinopril orally (PO), up-titrated to maximum tolerated doses as per standard clinical practice for 6 months.
  Interventions: Drug: Carvedilol; Drug: Lisinopril
- Group II (pravastatin, spironolactone) (Experimental): Patients receive standard clinical practice therapy as in Group I. Patients also receive pravastatin PO and spironolactone PO for 6 months.
  Interventions: Drug: Carvedilol; Drug: Lisinopril; Drug: Pravastatin; Drug: Spironolactone

INTERVENTIONS:
Drug: Carvedilol — Given PO
  Other Names: Coreg
Drug: Lisinopril — Given PO
  Other Names: N2-[(1S)-1-Carboxy-3-phenylpropyl]-L-lysyl-L-proline, Dihydrate; Prinivil; Zestril
Drug: Pravastatin — Given PO
  Other Names: [1S-[1alpha(betaS*,deltaS*),2alpha,6alpha,8beta(R*),8aalpha]]-1,2,6,7,8,8a-Hexahydro-beta,!d,6-trihydroxy-2-methyl-8-(2-methyl-1-oxobutoxy)-1-naphthaleneheptanoic Acid
  Arms: Group II (pravastatin, spironolactone)
Drug: Spironolactone — Given PO
  Other Names: 17-Hydroxy-7alpha-mercapto-3-oxo-17alpha-pregn-4-ene-21-carboxylic Acid, gamma Lactone, Acetate; Aldactone; SC 9420; SPL
  Arms: Group II (pravastatin, spironolactone)

SUMMARY:
This phase II trial compares two drug therapy plans for the correction of heart function changes (reduced ejection function) in patients who have undergone anthracycline-based treatment for lymphoma, sarcoma, or breast cancer. "Reduced ejection fraction" means the left ventricle of the heart is pumping a reduced blood volume with each heartbeat. Treatment is recommended, and the purpose of this research is to compare two different drug therapy plans (standard therapy with carvedilol and lisinopril and standard therapy with carvedilol and lisinopril plus pravastatin and spironolactone) and their effects on improvement of heart function. All of these drugs are heart medications, and carvedilol and lisinopril are commonly used to improve heart function. Adding pravastatin, a cholesterol lowering drug with additional beneficial effects on the cardiovascular system, and spironolactone, a water pill with additional beneficial effects on the cardiovascular system, may lead to even better (and faster) improvements in heart function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare cardiac function changes (delta left ventricular ejection fraction [LVEF]) over six months in patients with a new diagnosis of reduced LVEF after anthracycline-based therapy for lymphoma randomized to either standard therapy (carvedilol and lisinopril) or standard therapy plus pravastatin and spironolactone.

SECONDARY OBJECTIVE:

I. To compare cardiac function recovery rates over six months in patients with a new diagnosis of reduced LVEF after anthracycline-based therapy for lymphoma, sarcoma, or breast cancer randomized to either standard therapy (carvedilol and lisinopril) or standard therapy plus pravastatin and spironolactone.

II. To compare the time to recovery of cardiac function in patients with a new diagnosis of reduced LVEF after anthracycline-based therapy for lymphoma, sarcoma, or breast cancer randomized to either standard therapy (carvedilol and lisinopril) or standard therapy plus pravastatin and spironolactone.

OUTLINE: Patients are randomized in to 1 of 2 groups.

GROUP I: Patients receive carvedilol orally (PO) and lisinopril orally (PO), up-titrated to maximum tolerated doses as per standard clinical practice for 6 months.

GROUP II: Patients receive standard clinical practice therapy as in Group I. Patients also receive pravastatin PO and spironolactone PO for 6 months.

After completion of study treatment, patients are followed up at the 6 month visit.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age.
* New diagnosis of reduced cardiac function.
* Any prior anthracycline-based cancer therapy for hematological malignancy, breast cancer, or sarcoma.

Exclusion Criteria:

* History of heart failure (HF) of any class and type, or diagnosis of cardiomyopathy prior to anthracycline therapy.
* On active therapy with a fibrate, niacin or eplerenone, or statin.
* History of myopathy/rhabdomyolysis.
* History of statin intolerance.
* Active treatment for hyperlipidemia.
* History of gout.
* Active treatment for liver disease.
* Unexplained persistent elevations of serum transaminases (above upper limit of normal over two weeks).
* Pregnancy.
* Breast-feeding.
* Hyperkalemia (above upper limit of normal).
* Addison disease.
* Estimated glomerular filtration rate (eGFR) < 30 mL/minute/1.73 m^2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Delta change in left ventricular ejection fraction [LVEF]) | Baseline up to 6 months
  Will be a comparison of the average delta change in LVEF from start to six months of therapy between group 1 and 2 via an independent groups t-test or Wilcoxon as appropriate after testing distributional assumptions.

SECONDARY OUTCOMES:
Cardiac function recovery rates between group 1 and group 2 | Baseline up to 6 months
  Incidence rates will be compared using a simple test for equality of binomial proportions (χ ^ 2 -test or Fisher Exact).
Time to recovery of cardiac function between group 1 and group 2 | Baseline up to 6 months
  Will be a comparison of the average delta change in LVEF from start to six months of therapy between group 1 and 2 via an independent groups t-test or Wilcoxon as appropriate after testing distributional assumptions.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Herrmann, Principal Investigator — Mayo Clinic in Rochester